CLINICAL TRIAL: NCT05636449
Title: Ultrasound Guided Suprainguinal Fascia Iliaca Block vs. Periarticular Injection for Total Knee Arthroplasty: Prospective Randomized Study
Brief Title: Suprainguinal Fascia Iliaca Block vs. Periarticular Injection for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Oral Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ataunikneesurgery
Record Dates: First submitted 2022-11-15; First posted 2022-12-05 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Suprainguinal fascia iliaca block (Active Comparator): Suprainguinal fascia iliaca block after the surgery
  Interventions: Other: Group Suprainguinal fascia iliaca block
- Group Periarticular Infiltration Group (Active Comparator): A local anesthetic will be applied to the medial and lateral capsule, the medial and lateral meniscus margins, the deep part of the medial ligament, the medial and lateral synovial space, and the patellar ligament and quadriceps tendon.
  Interventions: Other: Group Periarticular Infiltration

INTERVENTIONS:
Other: Group Suprainguinal fascia iliaca block — After the operation is completed, the fascia iliaca will be separated from the iliacus muscle. With ultrasound guidance, the local anesthetic injection will be made between the fascia and the muscle.
  Arms: Group Suprainguinal fascia iliaca block
Other: Group Periarticular Infiltration — A total volume of 80 ml local anesthetic will be applied to the medial and lateral capsule, the medial and lateral meniscus margins, the deep part of the medial ligament, the medial and lateral synovial space, and the patellar ligament and quadriceps tendon.
  Arms: Group Periarticular Infiltration Group

SUMMARY:
Total knee replacement (total knee arthroplasty) is performed to resurface a knee damaged by arthritis and relieve pain in patients with severely damaged knee joints.

Total knee arthroplasty (TKA) is associated with severe postoperative pain, and the management of postoperative pain continues to evolve with the advancement of surgical techniques and pharmacological treatments.

Femoral, lateral femoral cutaneous nerve and obturator nerve block is provided with suprainguinal fascia iliaca plan block, which is used for postoperative analgesia, especially in hip surgeries. In this way, the investigators think it can be used as a part of multimodal analgesia in total knee arthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients
* Total knee arthroplasty

Exclusion Criteria:

* BMI>35
* liver, kidney, and advanced heart failure,
* routine use of analgesics and
* having used analgesics in the last 24 hours,
* having neuropathic pain,
* refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | first 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | first 48 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (between 0-10; 0: no pain, 10:worst pain) score
timed up and go test (TUG) | at 24th hour
  TUG- evaluation of the time in seconds for the patient to get up from the chair and walk 3 meters and return to the chair again
quadriceps muscle strength | at 24th hour
  will be evaluated in a scale between 1-5 (1:lowest; 5:normal)
joint range of motion test (ROM) | at 24th hour
  will be measured with goniometer( between 0-180 degrees)
Five Time Sit to Stand Test (FTSST) | at 24th hour
  physical assistance of the patient getting up and sitting down 'as fast as possible' five times without

CONTACTS AND LOCATIONS:
Overall Officials: Elif Oral Ahiskalioglu, Study Director — Ataturk University
Locations (1):
- Ali Ahiskalioglu, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suarez JC, Al-Mansoori AA, Kanwar S, Semien GA, Villa JM, McNamara CA, Patel PD. Effectiveness of Novel Adjuncts in Pain Management Following Total Knee Arthroplasty: A Randomized Clinical Trial. J Arthroplasty. 2018 Jul;33(7S):S136-S141. doi: 10.1016/j.arth.2018.02.088. Epub 2018 Mar 12. PMID 29628196
- [Background] Bravo D, Layera S, Aliste J, Jara A, Fernandez D, Barrientos C, Wulf R, Munoz G, Finlayson RJ, Tran Q. Lumbar plexus block versus suprainguinal fascia iliaca block for total hip arthroplasty: A single-blinded, randomized trial. J Clin Anesth. 2020 Nov;66:109907. doi: 10.1016/j.jclinane.2020.109907. Epub 2020 Jun 2. PMID 32502775